CLINICAL TRIAL: NCT01297101
Title: A National, Multi Center, Randomized, Open-label, Phase II Trial of Tarceva Versus Combination of Gemcitabine Plus Cisplatin as Neoadjuvant Treatment in Stage IIIA-N1,N2 NSCLC With Activating EGFR Mutation in Exon 19 or 21
Brief Title: Evaluating Efficacy and Safety of Erlotinib Versus Gemcitabine Plus Cisplatin as Neoadjuvant Chemotherapy
Status: Temporarily not available | Type: Expanded Access
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Lu Shun / Profess, Shanghai Chest Hospital
Other Study IDs: ML25268(C-TONG1101)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib — 150mg/qd, on day 15-28 of each 28 day cycle.
  Other Names: Tarceva

SUMMARY:
The aim of this study is to investigate the efficacy and safety of Tarceva versus combination of Gemcitabine plus Cisplatin as neoadjuvant treatment in patients with stage IIIA-N1,N2 NSCLC with EGFR activating mutation in exon 19 or 21.

DETAILED DESCRIPTION:
Concurrent Chemoradiation therapy remain the standard treatment for stage IIIA disease, but its treatment-related life threaten toxicity limit its use for those patients.

Tarceva monotherapy have been demonstrated a significant improvement in overall survival and disease progression free survival when used for the treatment of patients with metastatic NSCLC, after failure of at least one prior chemotherapy regimen. It is well tolerated without the side effects usually associated with chemotherapy.

Based on the encouraging results reported from the SLCG phase II study reported the efficacy of Tarceva as first line treatment for metastatic NSCLC with EGFR mutation patients would prolong overall survival, delay disease progression and be well tolerated, mOS reached 27 months, ORR reached 71%. Besides, with different mechanism and more tolerable than chemo, Tarceva may provide an important treatment alternative for local advanced pts with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed of non-small cell lung cancer
* Diagnosed as stage IIIA-NI, N2, except for T4N1M0
* The diagnosis standard of N1 or N2 is as below:
* The short axis of N1 lymph node of Stage IIIA-N1 must be ≥ 10 mm on Computed Tomography, and the Standard Uptake Value (SUV) on PET-CT of N1 lymph node must be > 2.5

Exclusion Criteria:

* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab)
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy)
* Resection of primary malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Chen Z, Shen S, Shi W, Jiang G, Wang X, Jian H, Zhou Z, Ding Z, Lu S. Intercalated combination of chemotherapy and erlotinib for stage IIIA non-small-cell lung cancer: a multicenter, open-label, single-arm, phase II study. Cancer Manag Res. 2019 Jul 12;11:6543-6552. doi: 10.2147/CMAR.S189287. eCollection 2019. PMID 31372055